CLINICAL TRIAL: NCT02653235
Title: Exploring the Impact of Peripheral Immune Challenge on the "Triple Network" and "Dorsal Nexus" Functional Connectivity in Humans
Brief Title: Impact of Immune Challenge on Triple Network Connectivity in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GN14NE490
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Typhoid vaccination (Active Comparator): Salmonella typhi vaccination
  Interventions: Biological: Salmonella typhi vaccination
- Placebo (Placebo Comparator): 0.9% sodium chloride
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Salmonella typhi vaccination
  Arms: Typhoid vaccination
Biological: Placebo
  Arms: Placebo

SUMMARY:
Acquiring, processing and utilising "information" is crucial to any mental function -including seemingly simple daily functions. Collectively called 'cognitive functions', these processes are a result of different regions of the brain acting together.

Disruption of these cognitive functions increases the risk of development of mental health problem. Recently it has been proposed that inflammatory pathways may contribute to disorders of cognition and behaviour like depression.

This is largely due to research showing that those with inflammatory conditions like arthritis are more likely to develop mental health problems like depression. Conversely, those who suffer from mental health problems (even in the absence of inflammatory conditions) have large amounts of inflammatory molecules in the blood. Studies in animals suggest that inflammation outside the brain can reach and affect the brain in a number of ways. So, does inflammation play a role in the development of cognitive and behavioural symptoms? What are the pathways involved?

The current project tries to address this question. Specifically, the investigators intend to use modern scanning techniques to examine the effect of inducing a low grade inflammation (using a commonly used typhoid vaccine) to see how the inflammation affects how different regions of the act together to perform cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 18 - 50 years old
3. Male

Exclusion Criteria:

1. Female
2. History/family history of medical or/and Axis I DSM IV condition
3. Received typhoid vaccination within the last 3 years
4. Taken oral antibiotics/antiinflammatory agents within the previous 2 weeks
5. Current Smokers
6. Contraindication for MRI scans
7. Contraindication for Salmonella typhi vaccination
8. Known hypersensitivity to a Vi antigen containing vaccine.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity measured using resting state functional MRI BOLD time series cross correlations between the network nodes. | 6 hours

SECONDARY OUTCOMES:
Correlation of functional connectivity measures with circulating serum cytokines and POMS/ BDI scores using multivariate general linear models | 6 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stefanov K, McLean J, McColl A, Basu N, Cavanagh J, Krishnadas R. Mild Inflammation in Healthy Males Induces Fatigue Mediated by Changes in Effective Connectivity Within the Insula. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Sep;5(9):865-874. doi: 10.1016/j.bpsc.2020.04.005. Epub 2020 Apr 22. PMID 32532687